CLINICAL TRIAL: NCT00471289
Title: Percutaneous Transluminal Balloon Angioplasty (PTA) and Drug Eluting Stents for Infrapopliteal Lesions in Critical Limb Ischemia
Brief Title: PTA and Drug Eluting Stents for Infrapopliteal Lesions in Critical Limb Ischemia
Acronym: PADI
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Netherlands Society for Interventional Radiology (Other)
Responsible Party: Principal Investigator, H. van Overhagen MD PhD, Radiologist Haga Teaching Hospital The Hague, Netherlands Society for Interventional Radiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PADI/200601
Record Dates: First submitted 2007-05-07; First posted 2007-05-09 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Peripheral Vascular Disease
Keywords: Critical Limb Ischemia; Stents; Drug Eluting Stents; Peripheral arterial disease; PAD; Paclitaxel; TAXUS; Infrapopliteal; Infragenicular; Interventional Radiology; CLI; DES
MeSH Terms: conditions — Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): PTA with primary placement of Drug (paclitaxel) Eluting Stent
  Interventions: Device: PTA with placement of paclitaxel-eluting stent
- 2 (Active Comparator): PTA
  Interventions: Device: PTA

INTERVENTIONS:
Device: PTA with placement of paclitaxel-eluting stent — PTA with placement of paclitaxel-eluting stent
  Arms: 1
Device: PTA — PTA
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the performance of paclitaxel-coated balloon expandable stainless steel coronary stent for the treatment of infrapopliteal stenoses and occlusions in patients with critical limb ischemia compared to percutaneous transluminal balloon angioplasty (PTA).

DETAILED DESCRIPTION:
Critical limb ischemia (CLI) is a serious condition that is becoming more and more common in the western world due to the growing percentage of elderly in the population and the rising incidence of diabetes. In about 40% of patients a stenosis or occlusion in the arteries below the level of the knee will be present. Restoration of blood flow is imperative to allow pain relief and tissue healing. Without revascularization patients with CLI are at risk for limb loss and potentially fatal complications such as sepsis.

In patients treated with percutaneous transluminal balloon angioplasty (PTA)significant restenosis is found in approximately 50% after 6 months.

In interventional cardiology a significant reduction in restenosis rates in coronary arteries has been found using drug eluting stents (DES), including the paclitaxel eluting stent (TAXUS, Boston Scientific). DES locally deliver drugs (e.g. paclitaxel) that interfere with the restenosis process.

Using DES in treating below the knee (infrapopliteal) arterial lesions in patients with CLI may improve patency and clinical outcome.

Comparison:

Treatment of below the knee arterial lesions in patients with CLI with PTA and DES compared to only PTA.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age > 18 years
* If female patient with child bearing potential, patient may not be pregnant at the study entry and must utilize reliable birth control for the duration of her participation into the study
* Patient is willing and able to comply with the specified follow-up evaluation
* Critical Limb Ischaemia, this is Fontaine stage III (ischaemic rest pain) and IV (ischaemic ulcers or gangrene) or Rutherford category 4 (ischaemic rest pain), 5 (minor tissue loss) or 6 (major tissue loss)
* Stenotic (>50% luminal loss) or occluded infrapopliteal artery, including the tibiofibular trunk, the anterior tibial artery, the posterior tibial artery and the peroneal artery, with a lesion length ≤ 60 mm
* Artery to be treated with a diameter more tham or equal to 2mm and less than or equal to 4mm
* Patent common iliac, external iliac, superficial femoral and popliteal artery on the ipsilateral side prior to randomisation, possibly after treatment during the same session
* At least one patent crural (anterior tibial, posterior tibial or peroneal) artery with expected unobstructed runoff to ankle level after treatment

Exclusion Criteria:

* Acute limb ischaemia
* Subacute limb ischaemia which requires thrombolysis as first treatment modality
* Active bleeding or bleeding diathesis
* Recent (less than 3 months) hemorrhagic stroke or other any other CNS abnormality with increased risk of haemorrhage, such as intracranial neoplasm, arteriovenous malformation, intracranial aneurysm or aneurysm repair
* Gastrointestinal or genitourinary bleeding of clinical significance within the previous 6 weeks before treatment
* Aneurysm in common femoral, superficial femoral or popliteal artery on the ipsilateral side
* Revascularization involving the same limb within 30 days prior to the index procedure or planned revascularization of the same limb within 30 days of the index procedure
* Previous implanted stent at the index site
* Life expectancy of less than 6 months or other factors making clinical follow-up difficult
* Known allergy to acetylsalicylic acid (aspirin), clopidogrel, heparin or paclitaxel
* Known allergy to contrast media
* Known heparin induced thrombocytopenia (HIT type 2)
* Patient unable or unwilling to tolerate anticoagulant, anti-platelet therapy or contrast media
* Creatinine clearance < 20 ml/min (as derived from Cockcroft-Gault or MDRD formula)unless patient is on hemodialysis
* Aneurysm in common femoral, superficial femoral or popliteal artery on the ipsilateral side
* Severely calcified lesions with expected resistance to stenting
* Poor inflow due to ipsilateral stenoses or occlusions of the iliac or femoropopliteal arteries that cannot be treated during the same session
* Significant vessel tortuosity or other parameters prohibiting access to the lesions and/or delivery of the stent
* Patients without (expected) distal runoff to the index site
* Previous implanted stent at the index site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2007-08; Primary Completion 2013-09 (Actual); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be primary patency of the treated site at 6 months. Primary patency is defined as <50% loss of luminal diameter at the treated site on CT arteriography (CTA) without re-intervention in the interim. | 6 months

SECONDARY OUTCOMES:
Primary patency of the treated sites at 3, 6 and 12 months after intervention assessed by duplex sonography (binary patency, <50% stenosis defined as PSV ratio <2.0) | 3, 6, 12 months
Clinical evaluation of the treated ischemic leg at 3, 6 and 12 months. | 3, 6, 12 months
Major amputation (at or above the ankle) of the trial leg at 3, 6 and 12 months | 3, 6, 12 months
Minor amputation (below the ankle excluding the toes) of the trial leg at 3, 6 and 12 months. | 3, 6, 12 months
Infrapopliteal surgical bypass of the trial leg at 3, 6 and 12 months. | 3, 6, 12 months
Infrapopliteal endovascular re-intervention of the trial leg at 3, 6 and 12 months. | 3, 6, 12 months
Peri-procedural (within 30 days) complications. | 30 days
Death. | 3, 6, 12 months
Clinical assessment primarily by Rutherford score for peripheral arterial disease | 2, 3, 4 and 5 years after treatment
  Clinical assessment outpatient clinic
Target lesion patency by means of duplex sonography | 2, 3, 4 and 5 years after treatment
  During outpatient clinic visits
Major amputation (at or above the ankle) of treated limb | yearly up to 10 years after treatment
  Assessment up to 5 years after treatment during outpatient clinic visits From 5 to 10 years by means of yearly evaluation of patient charts
Minor amputation (below the ankle excluding the toes) of the trial leg at 3, 6 and 12 months. | yearly up to 10 years after treatment
  From 2 to 5 years during outpatient clinic visits From 5 to 10 years yearly evaluation of patient charts
Endovascular or surgical re-intervention of target lesion | 3, 6, 12 months, 2,3,4 and 5 years after inclusion
  Follow-up until first re-intervention of target lesion

CONTACTS AND LOCATIONS:
Overall Officials: Hans Van Overhagen, MD PhD, Principal Investigator — HagaZiekenhuis Dept. of Radiology
Locations (3):
- Netherlands (3):
  - HagaZiekenhuis, location Leyweg, The Hague, South Holland
  - Sint Antonius Ziekenhuis, Nieuwegein, Utrecht
  - University Medical Center Utrecht (UMCU), Utrecht

REFERENCES:
- [Background] Management of peripheral arterial disease (PAD). TransAtlantic Inter-Society Consensus (TASC). Section D: chronic critical limb ischaemia. Eur J Vasc Endovasc Surg. 2000 Jun;19 Suppl A:S144-243. No abstract available. PMID 10957907
- [Background] Adam DJ, Beard JD, Cleveland T, Bell J, Bradbury AW, Forbes JF, Fowkes FG, Gillepsie I, Ruckley CV, Raab G, Storkey H; BASIL trial participants. Bypass versus angioplasty in severe ischaemia of the leg (BASIL): multicentre, randomised controlled trial. Lancet. 2005 Dec 3;366(9501):1925-34. doi: 10.1016/S0140-6736(05)67704-5. PMID 16325694
- [Background] Jensen SA, Vatten LJ, Myhre HO. The prevalence of chronic critical lower limb ischaemia in a population of 20,000 subjects 40-69 years of age. Eur J Vasc Endovasc Surg. 2006 Jul;32(1):60-5. doi: 10.1016/j.ejvs.2005.12.022. Epub 2006 Mar 2. PMID 16513377
- [Background] Black JH 3rd, LaMuraglia GM, Kwolek CJ, Brewster DC, Watkins MT, Cambria RP. Contemporary results of angioplasty-based infrainguinal percutaneous interventions. J Vasc Surg. 2005 Nov;42(5):932-9. doi: 10.1016/j.jvs.2005.06.024. PMID 16275450
- [Background] Sigala F, Menenakos Ch, Sigalas P, Baunach Ch, Langer S, Papalambros E, Hepp W. Transluminal angioplasty of isolated crural arterial lesions in diabetics with critical limb ischemia. Vasa. 2005 Aug;34(3):186-91. doi: 10.1024/0301-1526.34.3.186. PMID 16184838
- [Background] Hynes N, Mahendran B, Manning B, Andrews E, Courtney D, Sultan S. The influence of subintimal angioplasty on level of amputation and limb salvage rates in lower limb critical ischaemia: a 15-year experience. Eur J Vasc Endovasc Surg. 2005 Sep;30(3):291-9. doi: 10.1016/j.ejvs.2005.04.020. PMID 15939635
- [Background] Eskelinen E, Alback A, Roth WD, Lappalainen K, Keto P, Railo M, Eskelinen A, Lepantalo M. Infra-inguinal percutaneous transluminal angioplasty for limb salvage: a retrospective analysis in a single center. Acta Radiol. 2005 Apr;46(2):155-62. doi: 10.1080/02841850510022705. PMID 15902890
- [Background] Kudo T, Chandra FA, Ahn SS. The effectiveness of percutaneous transluminal angioplasty for the treatment of critical limb ischemia: a 10-year experience. J Vasc Surg. 2005 Mar;41(3):423-35; discussion 435. doi: 10.1016/j.jvs.2004.11.041. PMID 15838475
- [Background] Atar E, Siegel Y, Avrahami R, Bartal G, Bachar GN, Belenky A. Balloon angioplasty of popliteal and crural arteries in elderly with critical chronic limb ischemia. Eur J Radiol. 2005 Feb;53(2):287-92. doi: 10.1016/j.ejrad.2004.02.016. PMID 15664294
- [Background] Tsetis D, Belli AM. The role of infrapopliteal angioplasty. Br J Radiol. 2004 Dec;77(924):1007-15. doi: 10.1259/bjr/97382129. PMID 15569642
- [Background] Matsagas MI, Rivera MA, Tran T, Mitchell A, Robless P, Davies AH, Geroulakos G. Clinical outcome following infra-inguinal percutaneous transluminal angioplasty for critical limb ischemia. Cardiovasc Intervent Radiol. 2003 May-Jun;26(3):251-5. doi: 10.1007/s00270-003-0007-z. PMID 14562973
- [Background] Molloy KJ, Nasim A, London NJ, Naylor AR, Bell PR, Fishwick G, Bolia A, Thompson MM. Percutaneous transluminal angioplasty in the treatment of critical limb ischemia. J Endovasc Ther. 2003 Apr;10(2):298-303. doi: 10.1177/152660280301000220. PMID 12877613
- [Background] Haider SN, Kavanagh EG, Forlee M, Colgan MP, Madhavan P, Moore DJ, Shanik GD. Two-year outcome with preferential use of infrainguinal angioplasty for critical ischemia. J Vasc Surg. 2006 Mar;43(3):504-512. doi: 10.1016/j.jvs.2005.11.016. PMID 16520164
- [Background] Wiskirchen J, Schober W, Schart N, Kehlbach R, Wersebe A, Tepe G, Claussen CD, Duda SH. The effects of paclitaxel on the three phases of restenosis: smooth muscle cell proliferation, migration, and matrix formation: an in vitro study. Invest Radiol. 2004 Sep;39(9):565-71. doi: 10.1097/01.rli.0000133815.22434.55. PMID 15308939
- [Background] Serruys PW, Kutryk MJ, Ong AT. Coronary-artery stents. N Engl J Med. 2006 Feb 2;354(5):483-95. doi: 10.1056/NEJMra051091. No abstract available. PMID 16452560
- [Background] Aoki J, Colombo A, Dudek D, Banning AP, Drzewiecki J, Zmudka K, Schiele F, Russell ME, Koglin J, Serruys PW; TAXUS II Study Group. Peristent remodeling and neointimal suppression 2 years after polymer-based, paclitaxel-eluting stent implantation: insights from serial intravascular ultrasound analysis in the TAXUS II study. Circulation. 2005 Dec 20;112(25):3876-83. doi: 10.1161/CIRCULATIONAHA.105.558601. Epub 2005 Dec 12. PMID 16344384
- [Derived] Spreen MI, Martens JM, Knippenberg B, van Dijk LC, de Vries JPM, Vos JA, de Borst GJ, Vonken EPA, Bijlstra OD, Wever JJ, Statius van Eps RG, Mali WPTM, van Overhagen H. Long-Term Follow-up of the PADI Trial: Percutaneous Transluminal Angioplasty Versus Drug-Eluting Stents for Infrapopliteal Lesions in Critical Limb Ischemia. J Am Heart Assoc. 2017 Apr 14;6(4):e004877. doi: 10.1161/JAHA.116.004877. PMID 28411244
- [Derived] Spreen MI, Martens JM, Hansen BE, Knippenberg B, Verhey E, van Dijk LC, de Vries JP, Vos JA, de Borst GJ, Vonken EJ, Wever JJ, Statius van Eps RG, Mali WP, van Overhagen H. Percutaneous Transluminal Angioplasty and Drug-Eluting Stents for Infrapopliteal Lesions in Critical Limb Ischemia (PADI) Trial. Circ Cardiovasc Interv. 2016 Feb;9(2):e002376. doi: 10.1161/CIRCINTERVENTIONS.114.002376. PMID 26861113
- [Derived] Martens JM, Knippenberg B, Vos JA, de Vries JP, Hansen BE, van Overhagen H; PADI Trial Group. Update on PADI trial: percutaneous transluminal angioplasty and drug-eluting stents for infrapopliteal lesions in critical limb ischemia. J Vasc Surg. 2009 Sep;50(3):687-9. doi: 10.1016/j.jvs.2009.04.073. PMID 19700099